CLINICAL TRIAL: NCT03345264
Title: The Find Your PATHS (Pragmatic Assessment of a Tool to Help Survivors) to Sexual Health and Parenthood Study
Acronym: PATHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Cancer Society, Inc. (Other)
Collaborators: Will2Love, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PATHS IRB1094101
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cancer-related Problem/Condition; Sexuality; Fertility
Keywords: Sexual Dysfunction; Fertility Disorders; Cancer
MeSH Terms: conditions — Sexuality; Sexual Dysfunction, Physiological; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients, survivors, and partners (Experimental)
  Interventions: Behavioral: Online, interactive self-help program

INTERVENTIONS:
Behavioral: Online, interactive self-help program — Participants will receive access to the program, which provides: In-depth information specific to cancer sites and treatments, guidance on medical options for cancer-related sex or fertility problems, personalized goal-setting with progress tracking and relapse prevention, self-help exercises on overcoming sexual, relationship, and dating problems, videos of survivors' stories, and video vignettes with actors.

SUMMARY:
Concerns with sexual health and fertility are common among cancer patients, survivors and their partners. Literature reviews suggest that over 60% of survivors have reproductive health problems yet fewer than 20% get professional help. This study will test the uptake, use and effectiveness of online, interactive self-help programs for men and women with cancer. Participants in the study will receive up to 6 months of access to the self-help programs without charge. Navigation through the programs can be personalized by setting goals and following links to the most relevant information. The programs cover all cancer sites and common treatments, explaining sexual and fertility side effects. Programs also include step-by-step cognitive behavioral self-help exercises, guidance on available medical treatment options, decision aids, and video stories with actual survivors as well as vignettes with actors. Information for same-sex couples is included. Programs include suggestions on how partners can work together to cope with sexual or fertility issues.

The primary hypothesis is that participants will report improvements in sexual function and satisfaction from baseline to 3-month follow-up. Secondary hypotheses will investigate whether more extensive use of the program is associated with better outcomes (dose-response effect) and whether the intervention also improves secondary outcomes such as anxiety, depression, relationship satisfaction, and seeking medical help. Analyses from the data will investigate how many people who are informed of the study decide to participate (uptake), as well as how often participants visit the program and which parts are used most. Both the male and female programs have previously been shown to help cancer survivors and partners in published clinical trials.

Participants will be encouraged to invite a sexual partner to join the study, but that will be optional. Partners will be able to be linked for statistical analysis through their unique study identification numbers. Participants' use of the websites will be electronically tracked and compared with questionnaire outcome measures. Outcome measures include online, self-report questionnaires completed at baseline and 3-month follow-up. At 6-month follow-up, participants will complete 2 online ratings of the helpfulness of the programs. Privacy and security are carefully protected. The entire website meets standards for HIPAA (Health Insurance Portability and Accountability Act). Questionnaires are identified with study numbers rather than names or email addresses. Once the study data are analyzed, the list linking participant identifying information (names, email) and study numbers will be destroyed. Any publications resulting from the study will discuss group data and will not contain any information that could be used to identify an individual participant.

ELIGIBILITY:
Inclusion Criteria:

* Has had a diagnosis of cancer or is the intimate partner of a cancer patient/survivor
* Has a concern or wants to learn more about cancer-related issues with sexuality or fertility
* Has a way to access the website and questionnaires on the internet

Exclusion Criteria:

* Younger than age 18
* Does not read and understand English well enough to use the website independently
* Does not live in the United States
* Potential participant has already subscribed to the male or female self-help program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
PROMIS® (Patient-Reported Outcomes Measurement Information System) Brief Sexual Profile v2 Male | Change from baseline to 3 months post consent
  Construct: Sexual function and satisfaction in men; Total Score Range: 0-33; Higher values represent a better outcome
PROMIS® (Patient-Reported Outcomes Measurement Information System) Brief Sexual Profile v2 Female | Change from baseline to 3 months post consent
  Construct: Sexual function and satisfaction in women; Total Score Range: 0-49; Higher values represent a better outcome

SECONDARY OUTCOMES:
PROMIS® (Patient-Reported Outcomes Measurement Information System) Brief Anxiety Scale | Change from baseline to 3 months post consent
  Construct: General anxiety level; Total Score Range: 0-16; Higher scores represent a worse outcome
PROMIS® (Patient-Reported Outcomes Measurement Information System) Brief Depression Scale | Change from baseline to 3 months post consent
  Construct: Depressed Mood; Total Score Range: 0-16; Higher scores represent a worse outcome
Abbreviated Dyadic Adjustment Scale-4 | Change from baseline to 3 months post consent
  Construct: Relationship happiness; Total Score Range: 0-21; Higher scores represent a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tenbroeck Smith, Principal Investigator — American Cancer Society, Inc.; Leslie Schover, Principal Investigator — Will2Love, LLC
Locations (1):
- Will2Love, LLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No